CLINICAL TRIAL: NCT01992913
Title: Integrated Cognitive Behavior Therapy to Improve Work Outcomes in Schizophrenia
Brief Title: Building Employment Skills Through Therapy for Veterans
Acronym: BESTVet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1157-R
Record Dates: First submitted 2013-11-01; First posted 2013-11-25 (Estimated); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Cognitive Behavioral Therapy; Cognition; Vocational Rehabilitation; Supported Employment; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- integrated CBT with computerized cognitive remediation (Experimental): integrated CBT with computerized cognitive remediation
  Interventions: Behavioral: integrated Cognitive Behavioral Therapy; Behavioral: Computerized cognitive remediation (CCR)
- Treatment As Usual (Other): Treatment As Usual
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: integrated Cognitive Behavioral Therapy — Novel CBT paradigm for schizophrenia/schizoaffective disorder
  Other Names: iCBT
  Arms: integrated CBT with computerized cognitive remediation
Other: Usual Care — The usual care that Veterans receive - not limited in scope (i.e., subjects may participate in any/all available treatments, outside the study condition)
  Other Names: UC
  Arms: Treatment As Usual
Behavioral: Computerized cognitive remediation (CCR) — Part of the iCBT paradigm, a four month block of bi-weekly computerized cognitive remediation using BrainHQ program.
  Other Names: CCR
  Arms: integrated CBT with computerized cognitive remediation

SUMMARY:
Schizophrenia/Schizoaffective Disorder is associated with serious problems with cognitive skills, social skills, and functional skills (like employment). There is a new form of cognitive behavioral therapy called integrated cognitive behavioral therapy (iCBT) that specifically addresses the cognitive, social, and functional deficits of schizophrenia/schizoaffective disorder. This study compared iCBT to the usual care (UC) that Veteran's receive. The investigators compared iCBT to UC in subjects with schizophrenia/schizoaffective disorder who are enrolled in a Supported Employment (SE) program, and evaluate whether iCBT is more helpful in improving job attainment, and other areas of functioning, both right after treatment, and 6 months after the end of treatment.

DETAILED DESCRIPTION:
The objective of the current study was to evaluate whether integrated cognitive behavior therapy (iCBT) can improve engagement and success in an existing Supported Employment (SE) program among the most functionally disabled patients with schizophrenia/schizoaffective disorder. The iCBT condition also included computerized cognitive remediation. The primary specific aim was to determine whether iCBT will significantly improve work outcomes at post-treatment to a greater extent than Usual Care (UC) in low functioning patients with schizophrenia/schizoaffective disorder who join the SE program. The secondary aims were to evaluate the whether iCBT will significantly improve work outcomes at 6 month follow-up relative to UC, and whether iCBT will improve functional outcomes post-treatment and at follow-up relative to UC in subjects who join the SE program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DSM-IV schizophrenia or schizoaffective disorder (SCID)
* Severe/extreme functional disability [World Health Organization Disability Assessment Scale (WHODAS) score > 50]
* Clinical stability (as per primary mental health provider)
* Receiving treatment at the Veterans Administration
* Minimal engagement in psychiatric rehabilitation services (just psychiatrist and therapist/case management in the last 6 months)
* Eligible for and willing to be enrolled in Supported Employment program
* Age 18 to 65
* Proficient in English
* Able to give informed consent

Exclusion Criteria:

* Neurologic disease or damage that would make the diagnosis of schizophrenia questionable
* Current opioid or stimulant dependence (SCID)
* Not appropriate due to safety concerns (based on risk assessment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-06-12 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Sayers, PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans receiving treatment for schizophrenia or schizoaffective disorder at the Corporal Michael Crescenz VA Medical Center in the Mental Health Clinic were offered the opportunity to participate in a research project meant to test whether a CBT group treatment that included cognitive remediation enhanced the employment outcomes of a standard Supported Employment program. Recruitment began 6/2015 and enrollment ended 7/2019.
Pre-assignment Details: Eighty-seven Veterans completed baseline assessment and met study criteria. Twenty Veterans subsequently withdrew or were administratively withdrawn for clinical reasons from further participation, prior to randomization. Six more Veterans in the first cohort who were to be randomized to the TAU group were assigned to the iCBT group to obtain sufficient participants for an initial therapy group (i.e., ten to twelve). This violated random assignment, thus were administratively withdrawn.
Groups:
- Integrated CBT With Computerized Cognitive Remediation: Integrated CBT with computerized cognitive remediation (iCBT)
  Integrated Cognitive Behavioral Therapy: Novel CBT group treatment for schizophrenia/schizoaffective disorder
  Computerized cognitive remediation (CCR): Part of the iCBT paradigm, a four month block of bi-weekly computerized cognitive remediation using BrainHQ program.
  Participants were also enrolled in a Supported Employment program to support job attainment and continuation, and any other treatments that were available to Veterans at the VA Medical Center.
- Treatment As Usual: Treatment As Usual (TAU)
  The usual care that Veterans receive - not limited in scope (i.e., subjects may participate in any/all available treatments, outside the study condition).
  Participants were also enrolled in a Supported Employment program to support job attainment and continuation.
Period: Baseline Assessment
Arm/Group | Integrated CBT With Computerized Cognitive Remediation | Treatment As Usual
Started | 37 | 30
Completed | 37 | 30
Not Completed | 0 | 0
Period: 6 Month Assessment
Arm/Group | Integrated CBT With Computerized Cognitive Remediation | Treatment As Usual
Started | 37 (no withdrawals, but not all participants were available for assessment) | 30 (no withdrawals, but not all participants were available for assessment)
Completed | 37 | 30
Not Completed | 0 | 0
Period: 12 Month Assessment
Arm/Group | Integrated CBT With Computerized Cognitive Remediation | Treatment As Usual
Started | 37 | 30
Completed | 37 (no withdrawals, but not all participants were available for assessment) | 30 (no withdrawals, but not all participants were available for assessment)
Not Completed | 0 | 0
Period: 18 Month Assessment
Arm/Group | Integrated CBT With Computerized Cognitive Remediation | Treatment As Usual
Started | 37 | 30
Completed | 37 (no withdrawals, but not all participants were available for assessment) | 30 (no withdrawals, but not all participants were available for assessment)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were Veterans with schizophrenia or schizoaffective disorder receiving clinical services in Behavioral Health of a large VA Medical Center. Participants indicated they were interested in receiving supportive employment services for assistance in job seeking and support in maintaining employment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated CBT With Computerized Cognitive Remediation | Treatment As Usual | Total
Number analyzed (Participants) | 37 | 30 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.9) | 51.3 (12.2) | 48.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 32 | 25 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black of African American | 25 | 26 | 51
  Race: More than one race | 1 | 1 | 2
  Race: Native American, Alaskan native | 2 | 0 | 2
  Race: Caucasian | 9 | 3 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Non-Hispanic ethnicity: Hispanic | 0 | 1 | 1
  Hispanic or Non-Hispanic ethnicity: NonHispanic | 37 | 29 | 66
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 30 | 67
Primary Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia | 31 | 22 | 53
  Schizoaffective disorder | 6 | 8 | 14
Marital status [Count of Participants; unit: Participants] — Self-reported marital status at the time of entry into the study
  Participants
    Never married | 18 | 15 | 33
    Currently married | 4 | 3 | 7
    Separated | 4 | 2 | 6
    Divorced | 10 | 8 | 18
    Widowed | 0 | 1 | 1
    Cohabitating | 1 | 1 | 2
Brief Negative Symptom Scale [Mean (Standard Deviation); unit: units on a scale] — The Brief Negative Symptom Scale total score has a possible range from 0 - 73, with higher scores indicating a higher level of negative symptoms associated with schizophrenia.
  units on a scale | 28.5 (12.2) | 28.7 (10.6) | 28.6 (11.4)
Scale for the Assessment of Positive Symptoms [Mean (Standard Deviation); unit: units on a scale] — The Scale for the Assessment of Positive Symptoms has a possible range from 0 - 170, with higher scores indicating higher levels of positive symptoms of schizophrenia.
  units on a scale | 27.6 (20.1) | 30.5 (14.3) | 28.9 (17.7)

OUTCOME MEASURES:

1. Primary Outcome: Workforce Participation Measure - Total Number of Jobs Attained
Description: Measure completed by the support employment specialist that evaluates participation in the workforce: Total number of jobs attained per group across the full length of the study (Baseline to 18 month follow-up, study end)
Time Frame: Baseline to post-treatment (18-months)
Measure: Mean (Standard Deviation); unit: Number of jobs attained
Groups:
- iCBT Group: Integrative Cognitive Behavioral Therapy group (experimental group)
- TAU Group: Treatment as Usual group (control group)
Arm/Group | iCBT Group | TAU Group
Number analyzed (Participants) | 37 | 30
Number of jobs attained
  Baseline | 0 (0) | 0 (0)
  18 month follow-up (study end) | 0.95 (1.2) | 0.43 (0.68)

2. Primary Outcome: Overall Job Attainment Proportion
Description: This is the proportion of participants, by group, that attained at least one job during the active portion of the study.
Time Frame: Study start through 18 months of the active portion of the study.
Population: Participants with diagnoses of schizophrenia or schizoaffective disorder seeking employment
Measure: Count of Participants; unit: Participants
Arm/Group | iCBT Group | TAU Group
Number analyzed (Participants) | 37 | 30
Participants
  No job attainment | 16 | 20
  At least one job attained | 21 | 10
Statistical Analysis 1: Comparison: iCBT Group vs TAU Group; We conducted a 2 X 2 chi-square analysis of differences in proportion; Test type: Superiority; p < .05, Fisher Exact — Fisher's exact Test, "right-sided probability" based on a directional hypothesis
Statistical Analysis 2: Comparison: iCBT Group vs TAU Group; Chis Sq: group (iCBT/TAU) X Job attained (Yes/No); Test type: Superiority; p < .06, Chi-squared; ChiSq = 3.6562, df = 1; Odds Ratio (OR) = 2.65, 95% CI 2-sided [0.97 to 7.13] — OR, iCBT / TAU in job attainment

3. Primary Outcome: Job Participant Composite-hours Worked
Description: This is a composite of hours work per week X number of weeks worked, in each assessment period.
Time Frame: Baseline to study intervention start point (ranging from 1-10 months), then at 6 months after intervention start, 12 months after intervention start, and then 18 months after intervention start.
Measure: Mean (Standard Deviation); unit: Hours worked
Arm/Group | iCBT Group | TAU Group
Number analyzed (Participants) | 37 | 30
Hours worked
  Baseline to intervention start point | 96.5 (361.1) | 25.3 (83.6)
  Intervention start to 6 mos. | 109.3 (228.8) | 27.0 (118.5)
  6-12 mos. | 110.8 (221.6) | 77.3 (169.3)
  12-18 mos. | 123.5 (245.8) | 133.4 (304.3)
Statistical Analysis 1: Comparison: iCBT Group vs TAU Group; Compare the groups on proportions in employment at the 6 month assessment points; Test type: Superiority — A mixed effects logistic regression model was conducted on a binary work variable, with a random intercept, using the baseline measure as a binary covariate; p < 0.33, Mixed Models Analysis; df (1, 30) for the group X assessment interaction, adjusting for baseline differences in hours worked at the start of the intervention; Odds Ratio, log = -.90, 95% CI 2-sided [-2.67 to .89], Standard Error of Mean 0.91
Statistical Analysis 2: Comparison: iCBT Group vs TAU Group; Compare the groups on proportions in employment at the 12 month assessment points; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < .54, Mixed Models Analysis; F (1, 130) = 1.0, p<0.37, for the group X assessment interaction, adjusting for baseline differences in hours worked at the start of the intervention; Odds Ratio, log = .52, 95% CI 2-sided [-1.14 to 2.19], Standard Error of Mean 0.85
Statistical Analysis 3: Comparison: iCBT Group vs TAU Group; Compare the groups on proportions in employment at the 18 month assessment point; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.71, Mixed Models Analysis; [statistical method as in outcome 3, analysis 2]; Odds Ratio, log = 0.31, 95% CI 2-sided [-1.32 to 1.73], Standard Error of Mean 0.83

4. Secondary Outcome: Work Behavior Inventory
Description: Measure completed by the supported employment specialist that evaluates work quality in an employment setting, based on the job supervisor's report, using the overall impression rating, ranging from 1 (consistently needing improvement) to 5 (consistently superior performance). Only the job supervisor's was used, rather than other options possible with the measure.
Time Frame: Baseline, mid-treatment (6-months), end of treatment (12-months), and post-treatment (18-months)
Population: Participants from both groups were very reluctant for the interventionists to obtain formal Work Behavior Inventory ratings from their employers. It was clear that insufficient data would be obtained and so efforts to complete it were abandoned. No data analysis was possible with this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iCBT Group | TAU Group
Number analyzed (Participants) | 1 | 0
units on a scale
  Baseline | 5.0 (0) |
  6 months | 4.0 (0) |
  12 months: number analyzed (Participants) | 0 | 0
  18 months: number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Specific Levels of Functioning (SLOF)
Description: This is measure designed to assess individual social, work, and interpersonal functioning of individuals with severe mental illness. The possible total score ranges from 30 - 150 with higher scores representing higher levels of functioning.
Time Frame: Baseline, mid-treatment (6-months), end of treatment (12-months), and post-treatment (18-months)
Population: The number of participants available for assessment at each time point varied due to the variability in willingness on the part of the participants to complete these interviews. Thus, data available at each time point for each group varied across time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCBT Group | TAU Group
Number analyzed (Participants) | 37 | 30
score on a scale
  Baseline | 128.0 (12.87) | 123.0 (19.33)
  6 months: number analyzed (Participants) | 23 | 19
  6 months | 125.3 (18.1) | 127.8 (10.9)
  12 months: number analyzed (Participants) | 22 | 17
  12 months | 127.8 (13.1) | 127.2 (16.3)
  18 months: number analyzed (Participants) | 19 | 20
  18 months | 127.9 (13.3) | 121.1 (18.7)
Statistical Analysis 1: Comparison: iCBT Group vs TAU Group; Test type: Superiority — This is mixed model analysis of the group X assessment interaction. This analysis is the test of mean differences in level of functioning at the baseline assessment; p < 0.19, Fisher Exact; df (1, 114); Mean Difference (Final Values) = -5.03, Standard Error of Mean 3.82
Statistical Analysis 2: Comparison: iCBT Group vs TAU Group; Test type: Superiority — This is mixed model analysis of the group X assessment interaction. This analysis is the test of mean differences in level of functioning at the 6 month assessment; p < 0.99, Fisher Exact; df (1, 114); Mean Difference (Final Values) = 0.03, Standard Error of Mean 4.42
Statistical Analysis 3: Comparison: iCBT Group vs TAU Group; Test type: Superiority — This is mixed model analysis of the group X assessment interaction. This analysis is the test of mean differences in level of functioning at the 12 month assessment; p < 0.94, Fisher Exact; df (1, 114); Mean Difference (Final Values) = -0.33, Standard Error of Mean 4.54
Statistical Analysis 4: Comparison: iCBT Group vs TAU Group; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.14, Fisher Exact; df (1, 114); Mean Difference (Final Values) = -6.67, Standard Error of Mean 4.52

ADVERSE EVENTS:
Time Frame: Adverse events were noted from study beginning (baseline) until the study end for the last participant. Adverse events were assessed, at minimum, at each major assessment point, from Baseline to intervention start, a period of time that varied across participants from 1 to 10 months, intervention start to the 6 month assessment, 6 months to 12 months assessments, and 12 months to 18 months assessment.
Description: Adverse events were also noted as reported by the Veteran or by clinicians in the medical record of the participants at times other than major assessments. Ongoing medical events not conceivably associated with the study's psychosocial intervention were not noted or reported by study staff, unless the event was accompanied by inpatient treatment or death. This included incarceration, which occurred in two instances for these significantly disordered participants.
Arm/Group | iCBT Group | TAU Group
All-Cause Mortality (participants affected / at risk) | 2/37 | 0/30
Serious Adverse Events (participants affected / at risk) | 12/37 | 9/30
Other Adverse Events (participants affected / at risk) | 0/37 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iCBT Group (N=37) | TAU Group (N=30)
Inpatient psychiatric hospitalization (Psychiatric disorders) | 12 (28) | 9 (23) — admission to a psychiatric unit for reasons of increased psychiatric symptoms, including substance abuse
Inpatient surgical hospitalization (Surgical and medical procedures) | 1 (1) | 1 (1) — Inpatient hospitalization for reasons of planned or unplanned surgical procedure
Dizziness (General disorders) | 2 (2) | 0 (0)
Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — Rectal bleeding
Observation (General disorders) | 1 (1) | 0 (0) — Admitted for observation due to fluid restriction
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Weakness in legs, unknown origin
Colonscopy (Gastrointestinal disorders) | 1 (1) | 0 (0) — Admitted for colonoscopy
Hand injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Admitted for hand injury
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
General Medical (Surgical and medical procedures) | 0 (0) | 2 (2) — Admitted for "general medical purposes"--no other information availably
UTI/blood infection (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Blood infection that began with a urinary tract infection

LIMITATIONS AND CAVEATS:
The population for which this study was designed were highly functionally impaired by serious psychiatric illness as an effort to improve employment outcomes in this vulnerable group. This led to significant problems with the ability for participants to respond to and complete requests for ongoing participation in study activities and assessments. The significant missing data was the result of these issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT01992913/Prot_SAP_000.pdf